CLINICAL TRIAL: NCT06469931
Title: Comparison of the Effectiveness of ESWT and Ozone Therapy in Patients With Carpal Tunnel Syndrome
Brief Title: Ozone Therapy in Patients With Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Head of Physiotherapy and Rehabilitation Department, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/06-40
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; ESWT; Ozone therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Range of Motion, Articular; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone therapy group (Experimental): In addition to range of motion exercises for wrist and hand and splinting, 3 sessions of ozone therapy will be applied once a week.
  Interventions: Other: range of motion exercises; Other: ozone therapy
- Extracorporeal shock wave therapy group (Experimental): Patients in this group will receive ESWT once a week for 3 consecutive weeks in addition to range of motion exercisess for wrist and hand and splinting.
  Interventions: Other: range of motion exercises; Device: Extracorporeal shock wave therapy

INTERVENTIONS:
Other: range of motion exercises — In addition to range of motion exercises for wrist and hand and splinting, 3 sessions of ozone therapy will be applied once a week.
Device: Extracorporeal shock wave therapy — Patients in this group will receive ESWT once a week for 3 consecutive weeks in addition to range of motion exercises for wrist and hand and splinting.
  Arms: Extracorporeal shock wave therapy group
Other: ozone therapy — ozone therapy
  Arms: Ozone therapy group

SUMMARY:
ESWT (Extracorporeal Shock Wave Therapy), which has been used in the treatment of musculoskeletal diseases in recent years, has come to the agenda as a new treatment method in Carpal Tunnel Syndrome. Although the effectiveness of ESWT, splinting and exercise applications in CTS patients is known in the literature, studies on the effectiveness of ozone therapy are limited. The aim of this study was to compare the efficacy of ozone therapy and ESWT applied in addition to splinting and exercise applications in patients diagnosed with CTS. The study will consist of 2 groups. In addition to exercise and splinting, 3 sessions of ozone therapy will be applied once a week to study group.Patients in the control group will receive ESWT once a week for 3 consecutive weeks in addition to exercise and splinting.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy resulting from compression of the median nerve at the wrist level. Various methods are applied in the conservative treatment of CTS. These include modification of daily life, splinting, physical therapy modalities and exercise methods. ESWT (Extracorporeal Shock Wave Therapy), which has been used in the treatment of musculoskeletal diseases in recent years, has come to the agenda as a new treatment method in Carpal Tunnel Syndrome. Ozone therapy has trophic effects, analgesic effects, antioxidant, immunomodulator, anti-inflammatory and antitumoral effects. Although the effectiveness of ESWT, splinting and exercise applications in CTS patients is known in the literature, studies on the effectiveness of ozone therapy are limited. The aim of this study was to compare the efficacy of ozone therapy and ESWT applied in addition to splinting and exercise applications in patients diagnosed with CTS. The study will consist of 2 groups. In addition to exercise and splinting, 3 sessions of ozone therapy will be applied once a week to study group.Patients in the control group will receive ESWT once a week for 3 consecutive weeks in addition to exercise and splinting. Ultrasonographic examinations of the median nerve cross-sectional area will be performed using a LOGIQ P5 (Healthcare Ultrasound, Korea) and a high frequency 7-12 MHz linear probe. A hand dynamometer will be used to assess the grip strength of the hand.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65 who have been complaining for at least 3 months
* Diagnosed with mild or moderate Carpal Tunnel Syndrome

Exclusion Criteria:

* Cervical disc herniation or radiculopathy,
* Brachial plexus lesion
* Previous hand or neck surgery
* Pregnancy,
* History of fracture at the wrist level
* Inflammatory rheumatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Median nerve cross-sectional area | 2 minutes
  Patients will be positioned seated facing the assessor, with the volar aspect of the wrist facing the air and at rest on a pillow. In the proximal carpal tunnel (at the level of the pisiform bone), the median nerve hyperechoic inner border line will be continuously traced and the transverse section surface area will be measured.

SECONDARY OUTCOMES:
Pain assesment | 1 minute
  On a 10 cm straight line with values 0 and 10 marked, the patient will be asked to place a mark according to the severity of the hand and/or wrist pain being studied

OTHER OUTCOMES:
Hand grip strength assessment | 5 minutes
  A hand dynamometer will be used to evaluate the grip strength of the hand. Double, triple and lateral grip will be evaluated using a pinchmeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No